CLINICAL TRIAL: NCT03971253
Title: Japan Post-Marketing Surveillance - Specified Drug Use-results Survey for Peficitinib to Assess Safety and Effectiveness in the Patients With Rheumatoid Arthritis
Brief Title: Japan Post-Marketing Surveillance for Peficitinib to Assess Safety and Effectiveness in the Patients With Rheumatoid Arthritis
Status: Recruiting | Type: Observational
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 015K-MA-3311
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Post-Marketing Surveillance; ASP015K; Smyraf; Rheumatoid arthritis (RA); Peficitinib
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — peficitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peficitinib: Participants will receive peficitinib once daily after meal.
  Interventions: Drug: Peficitinib

INTERVENTIONS:
Drug: Peficitinib — Oral
  Other Names: ASP015K; Smyraf

SUMMARY:
The objective of this study is to investigate the safety and effectiveness in routine clinical practice and actual clinical setting for all patients with rheumatoid arthritis (RA) treated with peficitinib.

DETAILED DESCRIPTION:
This is a mandatory Post-Marketing Surveillance (PMS) requested by Pharmaceuticals and Medical Devices Agency (PMDA) as a part of the Japan-Risk Management Plan (J-RMP).

ELIGIBILITY:
Inclusion Criteria:

* All patients with rheumatoid arthritis (RA) treated with peficitinib for the first time.

Exclusion Criteria:

* Not applicable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rheumatoid arthritis (RA) treated with peficitinib for the first time.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Safety assessed by frequency of adverse events (AEs) | Up to 52 weeks
  An AE is defined as any unwanted medical occurrence after drug administration and which does not necessarily have a causal relationship with the treatment.
Safety assessed by frequency of adverse drug reactions (ADRs) | Up to 52 weeks
  AEs whose relationship to the study drugs could not be ruled out is considered adverse drug reaction. AEs that fall under either "Probable" or "Possible" or "Unassessable" should be defined as "AEs whose relationship to the study drugs could not be ruled out."
Safety assessed by frequency of serious infections | Up to 156 weeks
  Serious infections include tuberculosis, pneumonia, pneumocystis pneumonia, ichorrhemia and opportunistic infection.
Safety assessed by frequency of malignancy | Up to 156 weeks
  Frequency of malignancy found after drug administration.
Safety assessed by frequency of events leading to death | Up to 156 weeks
  Any events leading to death will be reported as serious AEs.
Safety assessed by frequency of AEs of special interests | Up to 156 weeks
  AEs of special interests include neutrophil decrease, lymphocyte decrease, hemoglobin decrease, Herpes zoster, gastrointestinal perforation, interstitial pneumonia, reactivation of Hepatitis B virus, hepatic function disorder, venous thromboembolism, cardiovascular events, rhabdomyolysis and myopathy.
Safety assessed by frequency of serious adverse events (SAEs) | Up to 156 weeks
  An AE is considered "serious" if, in the view of either the investigator, it results in any of the following outcomes: death, life-threatening, persistent or significant disability/incapacity or substantial disruption, congenital anomaly or birth defect, hospitalization or prolongation of hospitalization, or medically important events.
Safety assessed by frequency of serious adverse drug reactions (SADRs) | Up to 156 weeks
  SAEs whose relationship to the study drugs could not be ruled out is considered serious ADR. SAEs that fall under either "Probable" or "Possible" or "Unassessable" should be defined as "SAEs whose relationship to the study drugs could not be ruled out."
Disease activity score (DAS28) - C-reactive protein (CRP) | Up to 52 weeks
  DAS28-CRP will be calculated using data from Tender Joint Count (TJC) (28 joints), Swollen Joint Count (SJC) (28 joints), C-reactive protein (CRP) and Subject's Global Assessment of Arthritis (SGA) with the formula; DAS28-CRP = 0.56√(TJC) + 0.28√(SJC) + 0.36 ln (CRP (mg/dL) x 10 + 1) + 0.014 x SGA (mm) + 0.96.
  DAS28-CRP exceeding 5.1 is considered high disease activity; exceeding 3.2 and not greater than 5.1, moderate disease activity; exceeding 2.6 and not greater than 3.2, low disease activity.
DAS28- erythrocyte sedimentation rate (ESR) score | Up to 52 weeks
  DAS28-ESR will be calculated using data from TJC (28 joints), SJC (28 joints), ESR and SGA with the formula; DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR (mm/h) + 0.014 x SGA (mm).
  DAS28-ESR exceeding 5.1 is considered high disease activity; exceeding 3.2 and not greater than 5.1, moderate disease activity; exceeding 2.6 and not greater than 3.2, low disease activity.
Simplified Disease Activity Index (SDAI) score | Up to 52 weeks
  SDAI score will be calculated with formula SDAI = TJC + SJC + SGA + Physician's Global Assessment of Arthritis (PGA) + CRP.
  SDAI score exceeding 26 is considered high disease activity; exceeding 11 and not greater than 26, moderate disease activity; exceeding 3.3 and not greater than 11, low disease activity.
Clinical Disease Activity Index (CDAI) score | Up to 52 weeks
  CDAI score will be calculated with formula CDAI = TJC + SJC + SGA + PGA. CDAI score exceeding 22 is considered high disease activity; exceeding 10 and not greater than 22, moderate disease activity; exceeding 2.8 and not greater than 10, low disease activity.
Tender Joint Count (TJC) (28 joints) | Up to 52 weeks
  The investigator/sub-investigator will examine the participant for tender joints, assessing the 28 joints and confirm the location of each tender joint.
Swollen Joint Count (SJC) (28 joints) | Up to 52 weeks
  The investigator/sub-investigator will examine the participants for swollen joints, assessing the 28 joints and confirm the location of the swollen joints.
Erythrocyte sedimentation rate (ESR) | Up to 52 weeks
  ESR will be recorded from blood samples collected.
C-reactive protein (CRP) | Up to 52 weeks
  CRP will be recorded from blood samples collected.
Subject's Global Assessment of Arthritis (SGA) (visual analog scale (VAS)) | Up to 52 weeks
  The participant assesses his/her own disease activity on a VAS of 0 - 100 mm, corresponding from 'no disease activity' to 'very severe disease activity', on the questionnaire form.
Physician's Global Assessment of Arthritis (PGA) (VAS) | Up to 52 weeks
  The investigator assesses participant's disease activity on a VAS of 0 - 100 mm, corresponding from 'no disease activity' to 'very severe disease activity', on the questionnaire form.
European League Against Rheumatism (EULAR) Response Criteria | Up to 52 weeks
  Based on DAS28 scores and changes in DAS28 scores before and after treatment with the study drug, EULAR Response Criteria categorize response to treatment as "No response", "Moderate response," or "Good response."
Percentage of participants achieving DAS28-CRP scores for remission | Up to 52 weeks
  Percentage of participants with DAS28 scores less than 2.6.
Percentage of participants achieving DAS28-ESR scores for remission | Up to 52 weeks
  Percentage of participants with DAS28 scores less than 2.6.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (47):
- Japan (47):
  - Site JP00023, Aichi
  - Site JP00005, Akita
  - Site JP00002, Aomori
  - Site JP00012, Chiba
  - Site JP00038, Ehime
  - Site JP00018, Fukui
  - Site JP00040, Fukuoka
  - Site JP00007, Fukushima
  - Site JP00021, Gifu
  - Site JP00010, Gunma
  - Site JP00034, Hiroshima
  - Site JP00001, Hokkaido
  - Site JP00028, Hyōgo
  - Site JP00008, Ibaraki
  - Site JP00017, Ishikawa
  - Site JP00037, Kagawa
  - Site JP00046, Kagoshima
  - Site JP00014, Kanagawa
  - Site JP00039, Kochi
  - Site JP00043, Kumamoto
  - Site JP00026, Kyoto
  - Site JP00024, Mie
  - Site JP00004, Miyagi
  - Site JP00045, Miyazaki
  - Site JP00020, Nagano
  - Site JP00042, Nagasaki
  - Site JP00029, Nara
  - Site JP00015, Niigata
  - Site JP00003, Numakunai
  - Site JP00033, Okayama
  - Site JP00047, Okinawa
  - Site JP00027, Osaka
  - Site JP00044, Ōita
  - Site JP00041, Saga
  - Site JP00011, Saitama
  - Site JP00025, Shiga
  - Site JP00032, Shimane
  - Site JP00022, Shizuoka
  - Site JP00009, Tochigi
  - Site JP00036, Tokushima
  - Site JP00013, Tokyo
  - Site JP00031, Tottori
  - Site JP00016, Toyama
  - Site JP00030, Wakayama
  - Site JP00006, Yamagata
  - Site JP00035, Yamaguchi
  - Site JP00019, Yamanashi

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.